CLINICAL TRIAL: NCT05483114
Title: Comparison of the Precision in the Position of Brackets With Two Indirect Bonding Materials: Polyvinylsiloxane and Thermal Glue. Split-mouth Randomized Clinical Trial.
Brief Title: Comparison of Precision in Brackets Position in Two Indirect Bonding Materials
Acronym: IDBmaterials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Maria Monica Zamora, Principal investigator, Fundación Universitaria CIEO
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: UniCIEO Indirect bonding
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Orthodontic Appliance Complication; Malocclusion
Keywords: indirect bonding
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized clinical trial study, with 15 participants.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A double-blind study will be carried out, where the patient and the operators who will record the results will be blinded. It is not possible to blind the clinician who performs the indirect bonding process. The processing of the registration of the linear measurements and the statistical advisor will be blinded, this will be done by means of codes for each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyvinylsiloxane (Active Comparator): Accuracy of indirect bonding of self-ligating brackets made with polyvinylsiloxane transfers
  Interventions: Procedure: Accuracy of indirect bonding of self-ligating brackets made with polyvinylsiloxane transfers
- Thermal glue (Active Comparator): Accuracy of indirect bonding of self-ligating brackets made with thermal glue transfers
  Interventions: Procedure: Accuracy of indirect bonding of self-ligating brackets made with thermal glue transfers

INTERVENTIONS:
Procedure: Accuracy of indirect bonding of self-ligating brackets made with polyvinylsiloxane transfers — The uppethat consists of positioning brackets on a study model and they will be extended to the patient's mouth. .r hemiarch of each patient will be randomly placed to be cemented with a transfer tray made of polyvinylsiloxane thermal glue, by means of the indirect technique
  Arms: Polyvinylsiloxane
Procedure: Accuracy of indirect bonding of self-ligating brackets made with thermal glue transfers — The uppethat consists of positioning brackets on a study model and they will be extended to the patient's mouth. .r hemiarch of each patient will be randomly placed to be cemented with a transfer tray made of polyvinylsiloxane thermal glue, by means of the indirect technique
  Arms: Thermal glue

SUMMARY:
Objective: To compare the cementation precision of self-ligating brackets between two indirect bonding materials: polyvinylsiloxane and thermal glue.

Methods: Split-mouth randomized clinical trial study, with 15 participants. The study will be divided into two groups, Group 1: Polyvinylsiloxane and Group 2: Thermal glue.

DETAILED DESCRIPTION:
Patients from the self-ligation clinic who meet the inclusion criteria will be invited to participate and sign the informed consent. For the cementation of the brackets in each patient, the upper arch (right and left) will be divided from the second premolar on the right side to the second premolar on the left side, randomly assigned, to be cemented with a polyvinylsiloxane transfer tray and the other with thermal glue (materials selected for the study).

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition with the presence of teeth 15-25 with
* Crowding in the upper arch according to Little's irregularity index,
* Teeth with healthy enamel (without hypoplasias, fluorosis, amelogenesis imperfecta),
* Fully erupted teeth

Exclusion Criteria:

* Absence of teeth selected for the study or that required premolar extractions before starting alignment and leveling
* Patients with rehabilitation such as crowns, veneers, fractured dentition, atypical morphology
* Teeth whose bracket loosens at the time of the procedure due to failure of the union
* Poor oral hygiene
* Patients with any significant displacement of the tooth that could prevent seating of the transfer tray
* Study models with bubbles.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-11-29 (Estimated)

PRIMARY OUTCOMES:
Linear mesio-distal position | 2 weeks
  It is the difference in the maximum Euclidean distance (two-dimensional plane) between a point mesial and distal of the bracket in the working model and in the patient's tooth.
Linear occlusal-gingival position | 2 weeks
  It is the difference in the maximum Euclidean distance (two-dimensional plane) between a point occlusal and gingival of the bracket in the working model and in the patient's tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Zamora, DDS, Principal Investigator — Fundacion universitaria CIEO - Unicieo

IPD SHARING:
Plan to Share IPD: No